CLINICAL TRIAL: NCT00771602
Title: A Randomized Trial of Rituximab vs Alemtuzumab vs Alemtuzumab + Rituximab as Consolidation Therapy for Patients With Chronic Lymphocytic Leukemia (CLL) With Evidence of Residual Disease Following Prior Chemo(Immuno)Therapy
Brief Title: Alemtuzumab + Rituximab Consolidation in CLL
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of accrual.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0767
Record Dates: First submitted 2008-10-10; First posted 2008-10-13 (Estimated); Results first posted 2011-04-29 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2015-05

CONDITIONS: Chronic Lymphocytic Leukemia; Leukemia
Keywords: Chronic Lymphocytic Leukemia; Leukemia; CLL; PLL; SLL; Rituximab; Rituxan; Alemtuzumab; Campath
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia | interventions — Rituximab; Alemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Rituximab (Experimental): Group 1: 375 mg/m^2 IV Rituximab Alone
  Interventions: Drug: Rituximab
- Alemtuzumab (Experimental): Group 2: 30 mg SQ Alemtuzumab Alone
  Interventions: Drug: Alemtuzumab
- Rituximab + Alemtuzumab (Experimental): Group 3: 375 mg/m^2 Rituximab + 30 mg SQ Alemtuzumab
  Interventions: Drug: Rituximab; Drug: Alemtuzumab

INTERVENTIONS:
Drug: Rituximab — 375 mg/m^2 by standard IV (intravenous) infusion on days 1, 8, 15, and 22 of weeks 1-4.
  Other Names: Rituxan®
  Arms: Rituximab; Rituximab + Alemtuzumab
Drug: Alemtuzumab — Dose escalation of 3, 10 and 30 mg subcutaneously (SQ) during week 1, followed by dose of 30 mg subcutaneously three times weekly (e.g. Monday-Wednesday - Friday) starting on week 2 for a total of 12 weeks (2-13).
  Other Names: Campath®; Campath-1H
  Arms: Alemtuzumab; Rituximab + Alemtuzumab

SUMMARY:
The goal of this clinical research study is to find out how well Campath (alemtuzumab), Rituxan (rituximab), or a combination of the 2 drugs may control Chronic Lymphocytic Leukemia (CLL) that is left after chemotherapy. The safety of these drugs will also be studied.

DETAILED DESCRIPTION:
Study Drugs:

Alemtuzumab and rituximab are both monoclonal antibodies. Monoclonal antibodies are proteins designed to attach to a protein on the surface of the leukemia cell. By attaching to the leukemia cell, monoclonal antibodies alert the immune system to target that cell and kill it.

Study Groups:

If you are found to be eligible to take part in this study, you will be randomly assigned (as in the roll of a dice) to 1 of 3 groups. Group 1 will receive rituximab alone. Group 2 will receive alemtuzumab alone. Group 3 will receive both drugs together.

At the beginning of the study, the chance of being assigned into any of the groups is about equal. However, once enough participants are on study and the response rate in each group is known, you will have a slightly better chance of being assigned to the group with the highest response rate.

Study Drug Administration:

Group 1:

If you are in Group 1, rituximab will be given through a needle in your vein 1 time a week for 4 weeks. The first time you receive rituximab, it will be given over about 4-6 hours. Depending on any side effects you may have, the later infusions may be given over about 2-4 hours.

Before each dose of rituximab, you will receive drugs such as benadryl (diphenhydramine), Tylenol (acetaminophen), and sometimes steroids (either by mouth or into your vein) to try and prevent and/or help control side effects such as fevers and chills.

To help prevent infections, you will take the antibiotic valacyclovir (or a similar drug). Valacyclovir is taken 1 time a day every day. Your doctor will describe this to you in more detail.

Group 2:

If you are in Group 2, alemtuzumab will be given as an injection under your skin 3 times a week for 13 weeks. You will have to come to the clinic for each dose, learn how to inject it yourself, or have someone else taught how to inject you.

To help prevent infections, you will take the antibiotic trimethoprin/sulfamethoxazole (SMX). Your doctor will tell you if you will take the tablet 2 times a day either 3 times a week (Monday, Wednesday, and Friday) or 2 times a week (Saturday and Sunday). You will also take either the antibiotic valganciclovir or valacyclovir. Valganciclovir tablets are taken 2 times every day. Valacyclovir is taken 1 time a day every day. You will continue to take the antibiotics for at least 3 months after your last dose of alemtuzumab.

Group 3:

If you are in Group 3, rituximab will be given through a needle in your vein 1 time a week for 4 weeks. The first time you receive the rituximab, it will be given over about 4-6 hours. Depending on any side effects you may have, the later infusions may be given over about 2-4 hours.

Alemtuzumab will be given as an injection under your skin 3 times a week for 13 weeks. You will have to come to the clinic for each dose, learn how to inject it yourself, or have someone else taught how to inject you.

Before each dose of rituximab, you will receive drugs such as benadryl (diphenhydramine), Tylenol (acetaminophen), and sometimes steroids (either by mouth or into your vein) to try and prevent and/or help control side effects.

To help prevent infections, you will take the antibiotic trimethoprin/sulfamethoxazole (SMX). Your doctor will tell you if you will take the tablet 2 times a day either 3 times a week (Monday, Wednesday, and Friday) or 2 times a week (Saturday and Sunday). You will also take either the antibiotic valganciclovir or valacyclovir. Valganciclovir tablets are taken 2 times every day. Valacyclovir is taken 1 time a day every day. You will continue to take the antibiotics for at least 3 months after your last dose of alemtuzumab.

Study Visits:

Every week while you are receiving therapy, blood (about 1 tablespoon) will be drawn for routine tests.

Six (6), 12, and 18 weeks (+/- 1 week) after you begin receiving the study drug(s) and then every 6 months (+/- 1 month) after that, you will have bone marrow biopsies and/or aspirates to check the status of the disease and to check for residual disease.

Every 6 months (+/- 3 months) after you have stopped receiving therapy, you will have a physical exam and blood (about 1 tablespoon) will be drawn for routine tests.

If you are in Group 2 or 3, during Week 3 and 6, blood (about 1 teaspoon) will be drawn to check for the cytomegalovirus (CMV) infection. This infection may occur in people with weakened immune systems.

If your doctor thinks it is necessary, you will have a chest x-ray and/or other scans.

Length of Study:

If you are in Group 1, you will take the study drug for up to 4 weeks. If you are in Groups 2 or 3, you will take the study drug(s) for up to 13 weeks. You will be taken off treatment early if you have intolerable side effects.

You will remain on study as long as the disease does not get worse.

This is an investigational study. Rituximab is FDA approved and commercially available for non-Hodgkin's lymphoma. However, it is not approved for the treatment of CLL.

Alemtuzumab is FDA approved and commercially available. It has been approved for the treatment of CLL when given by vein. It has not been approved to be given as an injection under the skin or for treatment after chemotherapy.

Up to 100 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

* Patients with CLL, CLL/prolymphocytic leukemia (PLL), or Small Lymphocytic Lymphoma (SLL) who have achieved an National Cancer Institute-Working Group (NCI-WG) nodular partial (nPR) or complete response (CR) with documentation of residual disease by MRD flow cytometry following chemotherapy or chemoimmunotherapy.
* Patients with CLL, CLL/PLL, or SLL who have achieved an NCI-WG partial response (PR) following prior chemotherapy or chemoimmunotherapy.
* Age >/=18 years.
* ECOG performance status </=2.
* Serum creatinine </= 2 mg/dL; serum total bilirubin </= 2 mg/dL; serum AST or ALT <4 x ULN.
* Signed informed consent.
* Male and female patients who are fertile agree to use an effective barrier method of birth control (ie, latex condom, diaphragm, cervical cap, etc.) to avoid pregnancy. Female patients of childbearing potential (non-childbearing is defined as >/= 1 year post-menopausal or surgically sterilized) need a negative serum or urine pregnancy test within 14 days of study enrollment.

Exclusion Criteria:

* Past history of anaphylaxis following exposure to rat or mouse derived complementarity determining region (CDR)-grafted humanized monoclonal antibodies.
* Hormonal therapy within 2 weeks prior to study start. Hormonal replacement therapy is permitted.
* Active Hepatitis B (at least one of the following markers positive: HBsAg, HBeAg, IgM anti-HBc, HBV DNA).
* Previous treatment with alemtuzumab plus rituximab in combination.
* Pregnant or nursing women.
* History of HIV infection.
* Active uncontrolled infection (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment).
* Less than 6 months from the completion of prior chemotherapy or chemoimmunotherapy. Completion of prior chemoimmunotherapy is defined as the last day of therapy of the respective treatment regimen.
* Symptomatic CNS disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2008-08; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Faderl, M.D., Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M.D. Anderson's Website — http://mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 08/13/08 through 01/26/10. All participants recruited at UT MD Anderson Cancer Center.
Pre-assignment Details: Study was closed early as result of low accrual.
Groups:
- Rituximab: Group 1: 375 mg/m^2 intravenous (IV) Rituximab Alone
- Alemtuzumab: Group 2: 30 mg subcutaneously (SQ) Alemtuzumab Alone
Period: Overall Study
Arm/Group | Rituximab | Alemtuzumab | Rituximab + Alemtuzumab
Started | 1 | 0 | 0
Completed | 1 | 0 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rituximab | Alemtuzumab | Rituximab + Alemtuzumab | Total
Number analyzed (Participants) | 1 | 0 | 0 | 1
Age, Categorical [Number; unit: years]
  <=18 years | 0 |  |  | 0
  Between 18 and 65 years | 1 |  |  | 1
  >=65 years | 0 |  |  | 0
Gender [Number; unit: participants]
  Female | 0 |  |  | 0
  Male | 1 |  |  | 1
Region of Enrollment [Number; unit: participants]
  United States | 1 |  |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Molecular Remissions at 52 Weeks
Description: Molecular Remissions (minimal residual disease (MRD) flow cytometry-negative) after monoclonal antibody consolidation therapy. Molecular remission is defined as resolution of all detectable disease below the limits of the MRD flow cytometry assay sensitivity.
Time Frame: 52 weeks
Population: No analysis available participant ineligible for evaluation; study terminated due to slow accrual.
Arm/Group | Rituximab | Alemtuzumab | Rituximab + Alemtuzumab
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Progression-free Survival
Description: Progression-free survival (PFS) is measured from date of trial entry until documented progression of disease or death from any cause.
Time Frame: 52 weeks or until disease progression
Reporting Status: Not Posted
Measure: Number; unit: months

3. Secondary Outcome: 52 Week Toxicity Rate
Description: The definition of toxicities include any >/= grade 3 non-hematologic toxicity, >/= grade 3 infection, and any symptomatic (i.e. febrile) documented CMV (cytomegalovirus) reactivation, according to NCI-WG definitions.
Time Frame: 52 weeks
Reporting Status: Not Posted
Measure: Number; unit: participants

ADVERSE EVENTS:
Time Frame: Adverse event collection during total treatment duration of 12 weeks; Overall study period: August 13, 2008 to January 26, 2010.
Arm/Group | Rituximab | Alemtuzumab | Rituximab + Alemtuzumab
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 1/1 | 0/0 | 0/0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rituximab (N=1) | Alemtuzumab (N=0) | Rituximab + Alemtuzumab (N=0)
Fever, Low Grade (General disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes